CLINICAL TRIAL: NCT01459029
Title: High Dose D-Serine as Adjuvant Treatment for Recent Onset Schizophrenia : A Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: High Dose D-Serine as Adjuvant Treatment for Recent Onset Schizophrenia
Acronym: SATROS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Herzog Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 043211- HMO-CTIL
Record Dates: First submitted 2011-10-09; First posted 2011-10-25 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; NMDA receptor; D-serine; Recent onset; Negative symptoms; Cognition
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- D-serine (Active Comparator): D-serine up to 6000 mg/day subject to tolerability
  Interventions: Drug: D-serine
- Control (Placebo Comparator): Treatment with inert capsules (placebo)
  Interventions: Drug: D-serine

INTERVENTIONS:
Drug: D-serine — Adjuvant treatment with D-serine up to 6000 mg/day vs. placebo

SUMMARY:
The purpose of this study is to compare efficacy and safety of add-on treatment with a moderately high dose of D-serine, an NMDA-glycine site agonist, in young, recent onset schizophrenia patients who suffer from significant symptoms despite treatment with antipsychotics.

DETAILED DESCRIPTION:
Background: Recent advances in understanding the neurobiology underlying schizophrenia have underscored a pivotal role for a specific receptor for the neurotransmitter glutamate, the NMDA receptor, whose function may be impaired in the disorder. Enhancing transmission at the NMDA receptor may therefore provide a novel mechanism for treating schizophrenia. Over the past decade clinical trials that included supplementation with different compounds enhancing transmission at the NMDA receptor have provided positive results, particularly with D-serine. However, none of these trials focused specifically on young patients with recent onset schizophrenia. In addition, the optimal D-serine dose was not determined, although a preliminary report suggested that higher doses than those used in most studies may provide additional benefit, without significant safety concerns or side effects. Also, the pro-cognitive effects of D-serine were not systematically analyzed, although preliminary data supports a potential role for D-serine in ameliorating the cognitive deficits found in schizophrenia.

Research Design: Over a two year period, 54 patients, male or female, aged 18-30 years who fulfill DSM-IV criteria for schizophrenia or schizoaffective disorder, will be entered into a 12 week, parallel group, double blind, randomized controlled trial assessing the efficacy of placebo vs. DSR (up to 6000 mg/day) augmentation to standard antipsychotic therapy. First episode patients, and patients treated with clozapine, will be randomized separately. Patients will be entered into the trial in accordance with strict inclusion and exclusion criteria after the nature of the study has been explained to them and they have given written informed consent. Clinical evaluations will be performed at baseline and then at regular intervals during the trial. In addition, neurocognitive evaluations, electrophysiological assessments and determination of amino acids levels will be conducted at the beginning and end of the study. Treatment emergent adverse effects will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30
* Diagnosis of schizophrenia/schizoaffective disorder
* Recent onset (up to five years since onset of positive symptoms)
* Stable dose antipsychotic treatment for at least 4 weeks
* Baseline PANSS total score of at least 70
* Baseline PANSS negative subscale score of at least 20
* Clinically stable (stable CGI score for two consecutive weeks)

Exclusion Criteria:

* Criteria for other DSM-IV Axis I diagnoses are met
* Lifetime history of alcohol or substance dependence
* Alcohol or substance abuse within the past year
* Judged clinically to be at suicidal or homicidal risk
* Female patients who are pregnant or lactating.
* Patients with known intolerance to D-serine treatment
* Patients treated with ECT within 12 weeks prior to study entry
* Patients treated with TMS within 4 weeks prior to study entry
* Patients suffering from an unstable and/or untreated medical disorder
* Patients suffering from renal or hepatic dysfunction

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Total Score of the Positive and Negative Syndrome Scale (PANSS) | Biweekly for 12 weeks

SECONDARY OUTCOMES:
Change from Baseline in the Composite T-score of the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Battery | 12 weeks
Change from Baseline in the Subscales of PANSS | Biweekly for 12 weeks
Change from Baseline in the Clinical Global Impressions (CGI) | Biweekly for 12 weeks
Change from Baseline in the Scale for the Assessment of Negative Symptoms (SANS) | Biweekly for 12 weeks
Change from Baseline in the Calgary Depression Scale for Schizophrenia (CDSS | Biweekly for 12 weeks
Change from Baseline in the Quality of Life Scale (QOL) | Biweekly for 12 weeks
Change from Baseline in the Simpson-Angus Extrapyramidal Rating Scale (SAS) | Biweekly for 12 weeks
Change from Baseline in the Abnormal Involuntary Movement Scale (AIMS) | Biweekly for 12 weeks
Change from Baseline in the Udvalg for Kliniske Undersgelser (UKU) Side Effect Rating Scale | Biweekly for 12 weeks
Change from Baseline in the Prepulse Inhibition (PPI) of Startle | 12 weeks
  Patients with schizophrenia and their relatives may exhibit deficits in this operational measure of sensorimotor gating
Amino Acid Serum Levels | 12 weeks
  Glutamate, Glycine, D-serine

CONTACTS AND LOCATIONS:
Overall Officials: Amit Lotan, MD, Principal Investigator — Hadassah Medical Organization; Bernard Lerer, MD, Study Director — Hadassah Medical Organization; Uriel Heresco-Levy, MD, Study Director — Ezrath Nashim - Herzog Memorial Hospital
Locations (2):
- Israel (2):
  - Ezrath Nashim - Herzog Memorial Hospital & Community Clinics, Jerusalem
  - Hadassah Medical Organization, Jerusalem